CLINICAL TRIAL: NCT06771193
Title: RETRACE Study - Retrospective Observational Study Evaluating Disease Characteristics and Treatment Landscape of High-risk Locally Advanced (LA) or Recurrent / Metastatic (R/M) Cervical Cancer in Italy
Brief Title: Study on Disease Characteristics and Treatment in Locally Advanced or Recurrent / Metastatic Cervical Cancer in Italy
Acronym: RETRACE
Status: Recruiting | Type: Observational
Sponsor: MSD Italia S.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS102062
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer; Locally Advanced Cervical Cancer; Recurrent Cervical Cancer; Metastatic Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Multicenter, Observational, Retrospective charts review. Observational study with descriptive purpose only. Retrospective data capture in consecutive patients diagnosed with CC who attended the Oncologic Clinics from Jan 2018 to Dec 2021 (using medical records, either electronic or not), inserted in eCRF and analyzed.

DETAILED DESCRIPTION:
This is a multicenter, observational, retrospective study. The primary aim of this trial is to describe patients and disease characteristics, as well as treatment pattern of locally advanced and recurrent/metastatic cervical cancer (R/M and LACC) in Italy, through a retrospective data capture, from January 2018 to December 2021.

Eligible cervical cancer patients will be identified by reviewing medical records and physician notes (paper or electronic).

Disease will be defined as follow:

* Locally advanced cervical cancer: a large tumour within the cervix (more than 4cm) or it has grown into the tissues around the cervix, but the cancer has not spread to other organs; usually includes stage 2B, 3 and 4A (FIGO staging)
* Recurrent cervical cancer: local tumour regrowth or development of distant metastasis discovered 6 months or more after complete regression of the treatment (26)
* Metastatic cervical cancer: cancer spreads beyond the pelvis to other parts of the body; usually defined as stage 4B (FIGO staging) Moreover, the patients' characteristics will be stratified as low risk and high risk for locally advanced cervical cancer and differences between their treatment partners will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patient (or their legally acceptable representatives) must have signed and dated the Informed Consent & Privacy Form (ICF)
* Age ≥18 years
* Diagnosis of a cervical cancer
* Locally advanced stage (not suitable for curative surgery) or recurrent or metastatic disease
* Any treatment received between January 2018 and December 2021 for advanced disease

Exclusion Criteria:

* Patients participating in a pharmacological clinical trial for the treatment of advanced disease
* Patients who participated in a clinical trial
* Patients who were administered with Pembrolizumab, Olaparib or Levantinib or medications from these class of drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who attend the Oncologic Clinics authorized to participate in the study, with a record of diagnosed cervical cancer, treated between January 2018 and December 2021, will be eligible for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients receiving each different treatment pattern of LA, recurrent, and metastatic CC (%) | Retrospective data capture from Jan 2018 to Dec 2021
  Baseline and demographic characteristics will be summarized by standard descriptive summaries using absolute frequencies and proportions (%).
The proportion of patient with recurrence or dead after treatment and remission (%) | Retrospective data capture from Jan 2018 to Dec 2021
  Baseline and demographic characteristics will be summarized by standard descriptive summaries using absolute frequencies and proportions (%).
Median time from remission to recurrence | Retrospective data capture from Jan 2018 to Dec 2021
  The study aim is to describe the time from curative intervention to recurrence (for patients who had a curative surgery).
  Time to recurrence will be calculated and represented using Kaplan-Meier curves and summarized using median with 95% confidence interval.
Number of lines of treatment | Retrospective data capture from Jan 2018 to Dec 2021
  The aim of this analysis is to describe patients' treatment patterns in LA or R/M Cervical Cancer considering the high heterogeneity of treatment options in clinical setting and the lack of real-world data in Italy.
The costs in terms of resources utilization associated to the different treatment patterns of LA, recurrent and metastatic CC | Retrospective data capture from Jan 2018 to Dec 2021
  Healthcare services for the present study include drug costs, general hospital costs (based on number of patient admissions and days of hospitalization, outpatients' visits, emergency access), specialist consultations and concomitant medications related to safety issue, radiological procedures, laboratory exams.

SECONDARY OUTCOMES:
The proportion of patients who undergone screening program (%) | Retrospective data capture from Jan 2018 to Dec 2021
  Baseline characteristics such as adherence to a screening program, HPV subtype, and PD-L1 expression will be summarized by standard descriptive summaries using absolute frequencies and proportions (%).
HPV subtype typization, if available | Retrospective data capture from Jan 2018 to Dec 2021
  Baseline characteristics such as adherence to a screening program, HPV subtype, and PD-L1 expression will be summarized by standard descriptive summaries using absolute frequencies and proportions (%).
History of HPV related lesions (CIN 2+ lesion) | Retrospective data capture from Jan 2018 to Dec 2021
  Baseline characteristics such as adherence to a screening program, HPV subtype, and PD-L1 expression will be summarized by standard descriptive summaries using absolute frequencies and proportions (%).
The proportion of patients with PD-L1 >1% and >50% (%) | Retrospective data capture from Jan 2018 to Dec 2021
  To describe the expression profile of PD-L1 (if available in archive pathology reports).
  Baseline characteristics such as adherence to a screening program, HPV subtype, and PD-L1 expression will be summarized by standard descriptive summaries using absolute frequencies and proportions (%).

CONTACTS AND LOCATIONS:
Locations (11):
- Italy (11):
  - Oncologia Medica Policlinico Sant'Orsola Malpighi, Bologna, Bologna
  - Ginecologia ed Ostetricia A.O. Cannizzaro, Catania, Catania
  - Oncologia Medica 1 IRCCS Ospedale Policlinico San Martino, Genova, Genova
  - Unità di Ginecologia Oncologica Medica IRCCS Ospedale San Raffaele, Milan, Milano
  - Unità Ostetricia, Ginecologia e Ginecologia Oncologica medica Humanitas San Pio X, Milan, Milano
  - Oncologia A.O.U. di Modena - Policlinico, Modena, Modena
  - U.O.S. Trattamenti Innovativi dell'utero Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale, Napoli, Napoli
  - UOC Oncologia Medica ed Ematologia Azienda Ospedaliera Universitaria Luigi Vanvitelli, Napoli, Napoli
  - IRCCS Centro di Riferimento Oncologico (CRO), Aviano, Pordenone
  - U.O.C. Ginecologia Oncologica Policlinico Agostino Gemelli, Roma, Roma
  - UOC Oncologia Medica Ospedale Dell'Angelo - Mestre Azienda USL3 Serenissima, Mestre, Venezia